CLINICAL TRIAL: NCT07140445
Title: Monitoring Neurocognitive Dysfunction and the Impact of Metabolism and Physical Capacity After Paediatric Haematopoietic Stem Cell Transplantation (Abbreviation: MindMe)
Brief Title: Monitoring Neurocognitive Dysfunction and the Impact of Metabolism and Physical Capacity After Paediatric HSCT
Acronym: MindMe
Status: Not yet recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Child Cancer Foundation (Other); Danish Cancer Society (Other); Danish Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Hilde Hylland Uhlving, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: MindMe
Record Dates: First submitted 2025-07-24; First posted 2025-08-24 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Stem Cell Transplant; Late Effect; Neurocognitive Dysfunction; Paediatric Patients; Metabolic Syndrome; Physical Capacity
MeSH Terms: conditions — Cognition Disorders; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — A buccal swap, plasma, serum and PBMC's will be biobanked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Today the overall survival of childhood cancers has increased to above 85%. This increase is partially caused by treatment with bone marrow transplantation. A bone marrow transplantation is an efficient treatment against high-risk leukemia, as well as other life-threatening immunological and hematological diseases. However, it is unfortunately also related to the risk of developing a long series of late effects during early adulthood, such as reduced muscle mass, cardiovascular disease and diabetes.

Some survivors of bone marrow transplantation in childhood also seem to experience changes in cognitive functions. These changes may be experienced as difficulties with concentration, forgetfulness, learning difficulties, and challenges in school or the labour market. Currently, the extent of cognitive changes following bone marrow transplantation in childhood is not fully understood, nor how it relates to other late effects, and what can be done to prevent cognitive impairment.

This research project will examine cognitive function in a group of survivors of bone marrow transplantation in childhood and find out whether there is a correlation between reduced cognitive function and the occurrence of other late effects, including metabolic changes and reduced physical capacity. It will also explore associations between cognitive function at late follow up and blood-based biomarkers of neurological damage and systemic inflammation at the time of transplantation to identify predictors of reduced cognitive function.

The goal of the study is to evaluate the level of cognitive functioning after bone marrow transplantation in childhood, see how it relates to other late effect and identify risk factors and biomarkers in the blood that can predict which patients are at risk of neurocognitive impairment. The results of this study will hopefully contribute to optimizing the prevention and treatment of cognitive impairments following bone marrow transplantation in childhood, thereby improving the quality of life for survivors of bone marrow transplantation in childhood.

ELIGIBILITY:
Inclusion Criteria:

* =/> 7 years of age
* treatment with HSCT in Denmark since 2010
* treatment with HSCT was before the age of 18 years
* ability to speak and understand Danish.

Exclusion Criteria:

* diagnosed with infantile autism before their HSCT
* Downs Syndrome

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants: All survivors of paediatric HSCT in Denmark who have undergone transplantation since 2010, being at least 2 years after HSCT, and at least 7 years of age on the day of assessment are eligible. All participants must be able to speak and understand Danish as well as to understand the research project, to give informed consent to participate. For participants younger than 18 years, where the parents will give consent, at least one parent must speak Danish. Thus, the inclusion criteria are: at least 7 years of age, treatment with HSCT in Denmark since 2010 before the age of 18 years, and ability to speak and understand Danish.
  Exclusion criteria: Participants who were diagnosed with infantile autism before their HSCT or have Downs Syndrome will be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Intelligence quotient | Day 1
  Scored on the clinical neurocognitive tests Wechler Intelligence Scale for Children Fifth edition (WISC-V ) for participants 7-16.9 years of age and Wechler Adult Intelligence Scale Fourth edition (WAIS-IV) for participants 17 years of age or older. Scaled scores range from 0-19, higher = better performance.
verbal reasoning | Day 1
  Scored on the clinical neurocognitive tests Wechler Intelligence Scale for Children Fifth edition (WISC-V ) for participants 7-16.9 years of age and Wechler Adult Intelligence Scale Fourth edition (WAIS-IV) for participants 17 years of age or older. Scaled scores range from 0-19, higher = better performance.
verbal learning | Day 1
  Assessed by a neuropsychologist using Test of Memory and Learning, second edition (TOMAL--2) and Rey Complex Figure Test and Recognition Trial (RCFT).
  TOMAL-2 scores are age-based scaled scores; higher scores reflect better verbal memory performance.
  Scores for RCFT range from 0-36 with higher scores reflecting better visual memory.
non-verbal reasoning | Day 1
  Scored on the clinical neurocognitive tests Wechler Intelligence Scale for Children Fifth edition (WISC-V ) for participants 7-16.9 years of age and Wechler Adult Intelligence Scale Fourth edition (WAIS-IV) for participants 17 years of age or older. Scaled scores range from 0-19, higher = better performance.
working memory | Day 1
  Scored on the clinical neurocognitive tests Wechler Intelligence Scale for Children Fifth edition (WISC-V ) for participants 7-16.9 years of age and Wechler Adult Intelligence Scale Fourth edition (WAIS-IV) for participants 17 years of age or older. Scaled scores range from 0-19, higher = better performance.
executive functioning | Day 1
  Assessed by a neuropsychologist using Delis-Kaplan Executive Function System (D-KEFS) trailmaking test and verbal fluency test. D-KEFS subtests yield age-based scaled scores. Higher scores indicate better executive functioning.
sustained attention | Day 1
  Assessed by a neuropsychologist using Conners' Continuous Performance Test 3rd Edition (CPT-3). The test evaluates attention-related performance in areas of inattentiveness, impulsivity, sustained attention, and vigilance. Scaled scores (t-scores) range from 0-100, higher = better performance.
processing speed | Day 1
  Scored on the clinical neurocognitive tests Wechler Intelligence Scale for Children Fifth edition (WISC-V ) for participants 7-16.9 years of age and Wechler Adult Intelligence Scale Fourth edition (WAIS-IV) for participants 17 years of age or older. Scaled scores range from 0-19, higher = better performance.
fine motor skills | Day 1
  Assessed by a neuropsychologist using Delis-Kaplan Executive Function System (D-KEFS) trailmaking test. D-KEFS subtests yield age-based scaled scores. Higher score indicates better fine motor skills

SECONDARY OUTCOMES:
Waist circumference | Day 1
  Waist circumference will be measured at the level of the superior border of the iliac crest, at the end of a normal expiration with a tape measure to the nearest 0.1 cm, as suggested by The US National Cholesterol Education Programme. Patients will be classified according to the American Heart Association/National Heart, Lung, and Blood Institute (AHA/NHLBI) criteria for Metabolic Syndrome as defined in the 2005 scientific statement (Grundy et al., 2005).
Triglycerides | Day 1
  Blood samples will be drawn from a cannula placed in an antecubital vein or a dorsal vein in the hand. Patients will be classified according to the American Heart Association/National Heart, Lung, and Blood Institute (AHA/NHLBI) criteria for Metabolic Syndrome as defined in the 2005 scientific statement (Grundy et al., 2005).
HDL-cholesterol | Day 1
  Blood samples will be drawn from a cannula placed in an antecubital vein or a dorsal vein in the hand. Patients will be classified according to the American Heart Association/National Heart, Lung, and Blood Institute (AHA/NHLBI) criteria for Metabolic Syndrome as defined in the 2005 scientific statement (Grundy et al., 2005).
Fasting glucose | Day 1
  Blood samples will be drawn from a cannula placed in an antecubital vein or a dorsal vein in the hand. Patients will be classified according to the American Heart Association/National Heart, Lung, and Blood Institute (AHA/NHLBI) criteria for Metabolic Syndrome as defined in the 2005 scientific statement (Grundy et al., 2005).
Blood pressure | Day 1
  Blood pressure will be measured on the upper arm while sitting in the suppine position, after 10 minutes of rest, with an automated blood pressure monitor. Blood pressure will be measured three times, or untill there is less than 10 mmHg difference between measurements. The final blood pressure will be a mean of the two last measurements. Patients will be classified according to the American Heart Association/National Heart, Lung, and Blood Institute (AHA/NHLBI) criteria for Metabolic Syndrome as defined in the 2005 scientific statement (Grundy et al., 2005).
Hip circumference | Day 1
  Measurement of hip circumference at the widest part of the buttocks with a tape measure, to the nearest 0.1 cm.
Test of lower extremity isometric knee extension strength | Day 1
  Test of lower extremity isometric knee extension strength: will be assessed by measuring the rate of force development, maximal isometric force, and dynamic force capacity using a special-build strength ergometer (Gym 2000®) with a dynamometer (US2A100 kg, Holtinger, Germany) and amplifier. Data is collected through an AD-card (100 HZ) with customized software (LabVIEW ®, National Instruments, Texas, USA). The participant will be seated during the test. The participant's thigh, pelvis, and torso will be securely strapped to minimize movement and isolate the knee extension muscles. For the isometric test, the participant will be instructed to push against the lever arm of the dynamometer as hard and as quickly as possible for a few seconds without any movement at the knee joint.
Handgrip strength | Day 1
  Handgrip strength will be measured while standing, with the elbow free from the body and flexed 90 degrees. Participants will press as hard as possible on a handheld dynamometer. Handgrip strength (kg) is measured twice for both arms and the highest result will be used in the analyses. Handgrip strength is a measure of strength in the underarm and correlate with overall physical impairment.
Muscle performance: Timed-up-and-go | Day 1
  Participants will sit on a chair with both feet flat on the ground. Subsequently, participants will be instructed to stand up, walk 3 meters, turn around, walk back, and sit down as fast as possible. Each participant will perform the test three consecutive times and the fastest test will be used for the analyses. The timed-up-and-go test depends on lower body muscular strength and balance and reflects a person's ability to move in an everyday setting.
Muscle performance: Sit-to-stand 30 sec. | Day 1
  Sit-to-Stand 30 sec: The participant sits on a chair allowing the participant to flex the legs at a 90 degree angle. The participant is instructed to stand up straight, and return to sitting, as many times as possible in 30 sec. The arms should be crossed in front of the body or hanging by the side. Number of repititions is the outcome.
Muscle performance: Sit-to-stand 60 sec. | Day 1
  Sit-to-Stand 60 sec: The participant sits on a chair allowing the participant to flex the legs at a 90 degree angle. The participant is instructed to stand up straight, and return to sitting, as many times as possible in 60 sec. The arms should be crossed in front of the body or hanging by the side. Number of repititions is the outcome.
Cardiorespiratory fitness | Day 1
  performed on an electrical-break ergometer bicycle (Lode Corival Pediatric or Monark Ergomedic 839 E) using a modified Godfrey protocol. The participant will be instructed to keep a steady pace (70-80 rpm), while the workload increases gradually with 10-25 watts pr. minute until exhaustion. Oxygen uptake (VO2), heart rate (HR), minute ventilation (VE), respiratory exchange ratio (RER), breathing frequency (BF), and tidal volume (TV) will be measured continuously during the test using a transportable a portable Cortex Metamax 3B wireless spirometry system (Cortex, Leipzig, Germany). The participant will breathe into a Hans Rudolph Valve (2-wat NRBV, Hans Rudolph Inc., Kansas City, MO, USA). Heart rate and oxygen saturation will be measured during the test. Furthermore, two objective criteria need to be fulfilled before the test is valid: 1) heart rate >85% of estimated maximal heart rate 2) respiratory exchange ratio (RER)>1.1. The primary outcome will be the peak oxygen uptake (V02max
Maximal leg extension power | Day 1
  Maximal leg extension power: maximal voluntary muscle force will be measured from both legs following a fixed protocol. Leg extensor power will be measured using an extension Power Rig (Nottingham Power Rig, Queen's Medical Centre Nottingham, NG7 2UH, United Kingdom), with subjects positioned with joint angles as if the participant was rising from a chair. Participants are carefully instructed to keep their hands across the chest and to not move the upper body while pushing. Verbal encouragement will be given to ensure maximal performance. The participants extend one leg as forcefully as possible, and the velocity of the flywheel is measured by an opto-switch and used to calculate average leg extensor power in the push. Dominant leg will be tested, a minimum of 5 attempts is carried out for each leg, however the participant continues until two attempts are lower than the maximum. The result is expressed in watt (W).
Pediatric Quality of Life Inventory (PedsQL™) 4.0 Generic Core Scales - Child and Parent Report | Day 1
  The PedsQL 4.0 Generic Core Scales assess health-related quality of life in children across four domains: physical functioning, emotional functioning, social functioning, and school functioning. The instrument uses a 5-point Likert scale (0 = never a problem; 4 = almost always a problem) - lower score meaning better outcome.
Pediatric Quality of Life Inventory (PedsQL™) Multidimensional Fatigue Scale - Child and Parent Report | Day 1
  The PedsQL Multidimensional Fatigue Scale assesses fatigue in children in three domains: general fatigue, sleep/rest fatigue, and cognitive fatigue. It uses the same 5-point Likert scale (0 = never a problem; 4 = almost always a problem) - lower score meaning better outcome.
Cognitive functioning measured by the PROMIS® Cognitive Function Short Form 8a - Self-Report | Day 1
  The PROMIS® Cognitive Function Short Form 8a is an 8-item self-report questionnaire assessing perceived cognitive functioning in the past 7 days. It evaluates aspects such as memory, mental clarity, and concentration. Each item is scored on a 5-point Likert scale ranging from 1 ("very often") to 5 ("never") - higher scores indicate better subjective cognitive functioning.
Physical activity measured by the PROMIS® Physical Activity Short Form 4a - Self-Report | Day 1
  The PROMIS® Physical Activity Short Form 4a is a 4-item self-report questionnaire that assesses the frequency and intensity of physical activity during the past 7 days. Items are rated on a 5-point Likert scale, with higher scores indicating higher levels of physical activity.
Emotional and behavioral functioning measured by the Strengths and Difficulties Questionnaire (SDQ) | Day 1
  The Strengths and Difficulties Questionnaire (SDQ) is a brief screening tool used to assess emotional and behavioral functioning. It consists of 25 items covering five subscales: Emotional Symptoms, Conduct Problems, Hyperactivity/Inattention, Peer Relationship Problems, and Prosocial Behavior. Each item is rated on a 3-point scale: "Not true" (0), "Somewhat true" (1), or "Certainly true" (2). A Total Difficulties Score (0-40) is calculated by summing four of the five subscales (excluding Prosocial Behavior), where higher scores indicate more emotional or behavioral difficulties. Higher Prosocial scores (0-10) indicate better social functioning.
  Age-appropriate versions of the SDQ will be used: parent- and self-report forms for children and adolescents, and self-report form for participants aged 18 years and older.
Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2) | Day 1
  The Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2), is a standardized questionnaire assessing executive functions in everyday settings through parent or teacher reports. The questionnaire consist of 63 items (rated 1= never, 2 = sometimes, 3 = always). Higher scores indicate greater executive dysfunction.
Attention-Deficit/Hyperactivity Disorder Rating Scale (ADHD-RS) score | Day 1
  The Attention-Deficit/Hyperactivity Disorder Rating Scale (ADHD-RS) is a standardized questionnaire used to assess the severity of ADHD symptoms based on parent or teacher reports. Scores are calculated using standardized methods and normed according to Danish age- and gender-specific normative data. The scale consists of items rated on a 4-point scale (0 = never or rarely 3 = very often). Higher scores indicate greater severity of ADHD symptoms.

OTHER OUTCOMES:
Hepatic fat and NAFDL stage | Day 1
  Amount of hepatic fat (%), as measured on a MRI scan of the liver with PDFF/liverlab.
Body composition: Fat mass | Day 1
  Body fat mass (%) will be analyzed on a whole-body DEXA scan
Body composition: Fat free mass | Day 1
  Fat free mass (%), as a surrogate measure of lean mass, will be analyzed on a whole-body DEXA scan
Body composition: Bone mineral density | Day 1
  Bone mineral density, will be analyzed on a whole-body DEXA scan. Z- and T-scores will be calculated.
Body mass index (BMI) | Day 1
  BMI will be calculated based on measurements of height and weight. To measure height the participants will stand up straight against a wall, in bare feet looking straight forward, and will be measured to the nearest 0.1 cm. Weight will be measured on an automated weight wearing only light indoor clothing with empty pockets and no shoes. BMI is calculated as wieght in kg diveded by height in meters squared.
Total-cholesterol | Day 1
  Will be analyzed in a plasma sample. Blood samples will be drawn from a cannula placed in an antecubital vein or a dorsal vein in the hand.
LDL-cholesterol | Day 1
  Will be analyzed in a plasma sample. Blood samples will be drawn from a cannula placed in an antecubital vein or a dorsal vein in the hand.
Plasma Concentration of IGF-1 and IGFBP-3 | Day 1
  Insulin-like growth factor 1 (IGF-1) and insulin-like growth factor binding protein 3 (IGFBP-3) will be analyzed in plasma samples. Blood will be drawn from a cannula placed in an antecubital vein or a dorsal vein in the hand.
Plasma Concentration of Thyroid Hormones (T3, T4) and Thyroid Stimulating Hormone (TSH) | Day 1
  Thyroid hormones, triiodothyronine (T3) and thyroxine (T4) as well as thyroid stimulating hormone (TSH) will be analyzed in a plasma sample. Blood samples will be drawn from a cannula placed in an antecubital vein or a dorsal vein in the hand.
Plasma Concentration of Sex Hormones and Related Biomarkers (Testosterone, Estrogen, FSH, LH, Inhibin, AMH, SHBG, Androgens, Estrogens) | Day 1
  Levels of sex hormones -including testosterone, estrogen, follicle-stimulating hormone (FSH), luteinizing hormone (LH), inhibin, anti-Müllerian hormone (AMH), sex hormone-binding globulin (SHBG), androgen group, and estrogen group-will be analyzed in plasma samples Blood samples will be drawn from a cannula placed in an antecubital vein or a dorsal vein in the hand.
Markers of Inflammation and Immune Status | Day 1
  Blood samples will be analyzed for inflammatory and immune system biomarkers including C-reactive protein (CRP), ferritin, immunoglobulin A (IgA), immunoglobulin G (IgG), immunoglobulin M (IgM), leukocyte count and differential, reticulocyte count, and platelet count. Standardized assays will be used to quantify these markers, which indicate systemic inflammation and immune response.
  Blood samples will be drawn from a cannula placed in an antecubital vein or a dorsal vein in the hand.
Oral glucose tolerance test: Glucose | Day 1
  Analyses of plasma glucose levels during a 2 hour oral glucose tolerance test. Blood samples will be drawn before and 30, 60, 90, 120 minutes after the intake of 75 g of glucose disolved in 250 ml of water.
Oral glucose tolerance test: Insulin | Day 1
  Analyses of plasma insulin levels during a 2 hour oral glucose tolerance test. Blood samples will be drawn before and 30, 60, 90, 120 minutes after the intake of 75 g of glucose disolved in 250 ml of water.
Oral glucose tolerance test: C-peptide | Day 1
  Analyses of plasma c-peptide levels during a 2 hour oral glucose tolerance test. Blood samples will be drawn before and 30, 60, 90, 120 minutes after the intake of 75 g of glucose disolved in 250 ml of water.
Oral glucose tolerance test: Insulinogenic Index | Day 1
  Based on glucose and insulin values from the OGTT the insulinogenic Index will be calculated, as a measure of beta-cell function. Blood samples will be drawn before and 30, 60, 90, 120 minutes after the intake of 75 g of glucose disolved in 250 ml of water.
Concentration of Neurological Damage Biomarkers (NfL, BDNF, and S100B) in Biobanked Blood Samples | Until the end of the study
  Biobanked blood samples collected at the time of transplantation from participants in the SCORE-study will be analyzed for concentrations of neurofilament light chain (NfL), brain-derived neurotrophic factor (BDNF), and S100 calcium-binding protein B (S100B). These biomarkers will be measured using standardized laboratory methods and reported in appropriate units, reflecting neurological damage or neuroprotection status.
Markers of Coagulation and Hematological Status | Day 1
  Blood samples will be analyzed for coagulation markers and hematological parameters including activated partial thromboplastin time (APTT), international normalized ratio (INR), coagulation factors II, VII, and X, hemoglobin concentration, hemoglobin A1c, and reticulocyte group counts. These measurements will be reported in standard clinical units and reflect coagulation function and hematologic health. Blood samples will be drawn from a cannula placed in an antecubital vein or a dorsal vein in the hand.
Tanner-stage | Day 1
  Tanner stage as assessed at clinical examination by a Medical Doctor. If the participant does not wish to undress the choice of subjectively assessing their own stage by looking at a poster of the different stages will be made.
VLDL-cholesterol | Day 1
  Will be analyzed in a plasma sample. Blood samples will be drawn from a cannula placed in an antecubital vein or a dorsal vein in the hand.
Markers of Liver and Kidney Function | Day 1
  Blood samples will be analyzed for biomarkers reflecting liver and kidney function, including alanine transaminase (ALAT), aspartate transaminase (ASAT), alkaline phosphatase, bilirubin, albumin, creatinine, urea (carbamid), calcium, phosphate, magnesium, sodium, potassium, and lactate dehydrogenase (LDH). Concentrations will be measured using standardized laboratory methods and reported in appropriate units. These markers reflect hepatic and renal functional status. Blood samples will be drawn from a cannula placed in an antecubital vein or a dorsal vein in the hand.
Vitamin and Mineral Levels | Day 1
  Plasma concentrations of vitamin D (25-Hydroxy-Vitamin D [D3+D2]) and essential minerals including calcium, magnesium, phosphate, sodium, and potassium will be measured using standardized laboratory methods. These markers provide information on nutritional and mineral balance status.
  Blood samples will be drawn from a cannula placed in an antecubital vein or a dorsal vein in the hand.
Chronic Graft-Versus-Host evaluation | Day 1
  Chronic Graft-Versus-Host Disease (cGVHD) presence and stage will be evaluated according to recommendations published by Jagasia et al 2015 (Doi: 10.1016/j.bbmt.2014.12.001)

CONTACTS AND LOCATIONS:
Overall Officials: Hilde H Uhlving, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Capital Region, Denmark